CLINICAL TRIAL: NCT00440167
Title: Randomized Phase III Trial With Capecitabine/Erlotinib Followed of Gemcitabine Versus Gemcitabine/Erlotinib Followed of Capecitabine in Patients With Advanced Pancreatic Cancer
Brief Title: Capecitabine/Erlotinib Followed of Gemcitabine Versus Gemcitabine/Erlotinib Followed of Capecitabine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PD Dr. med. Volker Heinemann (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, PD Dr. med. Volker Heinemann, Sponsor Delegatated Person, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RC-57 crossover
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Pancreatic Cancer
Keywords: capecitabine; gemcitabine; Erlotinib; pancreatic cancer; advanced
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Capecitabine; Erlotinib Hydrochloride

ARMS (2):
- Arm A (Active Comparator)
  Interventions: Drug: Capecitabine; Drug: Erlotinib
- Arm B (Active Comparator)
  Interventions: Drug: Gemcitabine; Drug: Erlotinib

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m², d 1, 8 , 15, q d28
  Arms: Arm B
Drug: Capecitabine — Capecitabine 2 x 1000 mg/m²/ d oral, d 1 - 14 followed by 7 days Pause ("Flat Dosing")
  Arms: Arm A
Drug: Erlotinib — Erlotinib 150 mg/d oral, daily without break

SUMMARY:
This crossover trial is performed in advanced and metastatic pancreatic cancer not previously exposed to chemotherapy. The study compares a standard arm with gemcitabine plus erlotinib to an experimental arm with capecitabine plus erlotinib. It is the first trial of its kind to incorporate second-line treatment into the study design. Patient who fail on first-line therapy are switched to the comparator chemotherapy without erlotinib. The trial therefore not only compares two different regimens of first-line treatment, it also compares two sequential treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Histologically proven pancreatic cancer stage III or IV (T1-3 N1M0 or T1 3N0 1M1)
* No option for resection with curative intent
* At least one measurable or not measurable lesion (according to RECIST)
* No previous chemotherapy or other systemic tumor therapy
* No previous radiation
* Performance-Status 0-2 according to WHO/ECOG
* Life expectancy of at least 3 months
* Adequate kidney-, liver- and bone marrow function, defined as
* Absolute neutrophil count * 1,5 x 109/l
* Hemoglobin * 8 g/dl
* Thrombocytes * 100 x 109/l
* Bilirubin * 2 x upper norm (with liver mets < 5-fold)
* Serum Creatinine * 1,25 x upper norm
* Creatinine clearance > 30 ml/min (Cockroft/Gault)
* Transaminases * 2,5 x upper norm (with liver mets < 5-fold)
* Possibility of regular long-term follow-up
* Negative pregnancy test in women at childbearing age
* All patients must have signed an informed consent before study entry.

Exclusion Criteria:

* Known secondary cancer other than curatively treated basalioma or carcinoma in situ of the cervix uteri
* Clinically unstable CNS-metastases
* Known hypersensitivity against study medication
* Severe impairment of renal function (creatinine clearance < 30 ml/min)
* Severe impairment of liver function (bilirubin > 2,0 x above upper norm, transaminases > 2,5 x upper norm, or with known liver metastasis >5 x upper norm)
* Clinically relevant disease of the cardiovascular system or other vital organs
* Known polyneuropathy
* Known DPD-deficiency (screening not required)
* Simultaneous treatment with the antiviral agent sorivudin or chemically related agents such as brivudin
* Pregnancy, lactation or lack of reliable contraception in women at childbearing age
* Mental disease, drug- or alcohol abuse
* Participation in another clinical trial within the last 4 weeks
* All other diseases which may prevent adequate participation in the trial
* Indication of lack of compliance with study regulations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2006-06; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
TTF2 | approximate 6 months after first line treatment
  Time to treatment failure, after 2nd line (crossover) therapy

SECONDARY OUTCOMES:
TTF1 | approximate 6 months after randomization
  Time to treatment failure
Remission Rate | approximate 6 months after randomization
Overall Survival | 42 months after randomization
Clinical Benefit Response | approximate 6 months after randomization
Tumor marker CA19-9 characteristics | approximate 6 months after randomization
Quality of Life | approximate 6 months after randomization
Toxicity | approximate 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, MD, Principal Investigator — University of Munich - Klinikum Grosshadern

REFERENCES:
- [Derived] Weiss L, Heinemann V, Fischer LE, Gieseler F, Hoehler T, Mayerle J, Quietzsch D, Reinacher-Schick A, Schenk M, Seipelt G, Siveke JT, Stahl M, Vehling-Kaiser U, Waldschmidt DT, Dorman K, Zhang D, Westphalen CB, von Bergwelt-Baildon M, Boeck S, Haas M. Three-month life expectancy as inclusion criterion for clinical trials in advanced pancreatic cancer: is it really a valid tool for patient selection? Clin Transl Oncol. 2024 May;26(5):1268-1272. doi: 10.1007/s12094-023-03323-1. Epub 2023 Oct 4. PMID 37794220
- [Derived] Guenther M, Surendran SA, Haas M, Heinemann V, von Bergwelt-Baildon M, Engel J, Werner J, Boeck S, Ormanns S. TPX2 expression as a negative predictor of gemcitabine efficacy in pancreatic cancer. Br J Cancer. 2023 Jul;129(1):175-182. doi: 10.1038/s41416-023-02295-x. Epub 2023 May 4. PMID 37142730
- [Derived] Guenther M, Haas M, Heinemann V, Kruger S, Westphalen CB, von Bergwelt-Baildon M, Mayerle J, Werner J, Kirchner T, Boeck S, Ormanns S. Bacterial lipopolysaccharide as negative predictor of gemcitabine efficacy in advanced pancreatic cancer - translational results from the AIO-PK0104 Phase 3 study. Br J Cancer. 2020 Oct;123(9):1370-1376. doi: 10.1038/s41416-020-01029-7. Epub 2020 Aug 24. PMID 32830200
- [Derived] Ormanns S, Siveke JT, Heinemann V, Haas M, Sipos B, Schlitter AM, Esposito I, Jung A, Laubender RP, Kruger S, Vehling-Kaiser U, Winkelmann C, Fischer von Weikersthal L, Clemens MR, Gauler TC, Marten A, Geissler M, Greten TF, Kirchner T, Boeck S. pERK, pAKT and p53 as tissue biomarkers in erlotinib-treated patients with advanced pancreatic cancer: a translational subgroup analysis from AIO-PK0104. BMC Cancer. 2014 Aug 28;14:624. doi: 10.1186/1471-2407-14-624. PMID 25164437
- [Derived] Heinemann V, Vehling-Kaiser U, Waldschmidt D, Kettner E, Marten A, Winkelmann C, Klein S, Kojouharoff G, Gauler TC, von Weikersthal LF, Clemens MR, Geissler M, Greten TF, Hegewisch-Becker S, Rubanov O, Baake G, Hohler T, Ko YD, Jung A, Neugebauer S, Boeck S. Gemcitabine plus erlotinib followed by capecitabine versus capecitabine plus erlotinib followed by gemcitabine in advanced pancreatic cancer: final results of a randomised phase 3 trial of the 'Arbeitsgemeinschaft Internistische Onkologie' (AIO-PK0104). Gut. 2013 May;62(5):751-9. doi: 10.1136/gutjnl-2012-302759. Epub 2012 Jul 7. PMID 22773551